CLINICAL TRIAL: NCT02223767
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Treatment of Height Phobics
Brief Title: TMS Augmented Exposure Therapy
Acronym: BEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Wuerzburg177/12; 098_MH (Other: Clinic for Psychiatry)
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Phobia
Keywords: TMS; virtual reality (VR); Exposure therapy; TMS augmentations of exposure therapy
MeSH Terms: conditions — Phobic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum transcranial magnetic stimulation (TMS) (Experimental): 10 Hz TMS over medial prefrontal cortex
  Interventions: Device: Experimental: Verum TMS
- Sham transcranial magnetic stimulation (TMS) (Experimental): 10 Hz sham TMS over medial prefrontal cortex
  Interventions: Device: Experimental: Sham TMS

INTERVENTIONS:
Device: Experimental: Verum TMS — Intensity of 100 % of the resting motor threshold with 10 Hz and intertrial interval (ITI) of 26 s. 1560 pulse in 40 trains at all . One train lasts 4 s.
  Arms: Verum transcranial magnetic stimulation (TMS)
Device: Experimental: Sham TMS — Sham stimulation with 10 Hz and ITI of 26 s. 1560 pulse in 40 trains at all . One train lasts 4 s.
  Arms: Sham transcranial magnetic stimulation (TMS)

SUMMARY:
This study investigates the beneficial effects of prefrontal brain stimulation (with a facilitating TMS protocol) before exposure therapy in acrophobic patients. The two exposure sessions were realized in virtual reality. Before and after therapy, the phobic symptoms were measured on a subjective, behavioral and physiological level. The placebo-controlled single blinded study includes 50 phobic patients, which were randomized into verum or sham TMS.

ELIGIBILITY:
Inclusion Criteria:

Criteria for a simple phobia: specific heights

Exclusion Criteria:

Objective tinnitus Involvement in psychiatric treatments Clinically relevant psychiatric comorbidity Clinically relevant unstable internal or neurological comorbidity History of or evidence of significant brain malformation or neoplasm, head injury Cerebral vascular events Neurodegenerative disorder affecting the brain or prior brain surgery Metal objects in and around body that can not be removed Pregnancy Alcohol or drug abuse history of seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Herrmann, PhD, Principal Investigator — University of Würzburg
Locations (1):
- University hospital, Würzburg, Germany

REFERENCES:
- See also: Related Info — http://www.ppp.ukw.de/beat

RESULTS

PARTICIPANT FLOW:
Groups:
- Verum TMS: 10 Hz transcranial magnetic stimulation (TMS) over medial prefrontal cortex
  Experimental: Verum TMS: Intensity of 100 % of the resting motor threshold with 10 Hz and intertrial interval (ITI) of 26 s. 1560 pulse in 40 trains at all . One train lasts 4 s.
- Sham TMS: 10 Hz sham TMS over medial prefrontal cortex
  Experimental: Sham TMS: Sham stimulation with 10 Hz and ITI of 26 s. 1560 pulse in 40 trains at all . One train lasts 4 s.
Period: Overall Study
Arm/Group | Verum TMS | Sham TMS
Started | 24 | 23
Completed | 20 | 19
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Verum TMS: 10 Hz TMS over medial prefrontal cortex
  Experimental: Verum TMS: Intensity of 100 % of the resting motor threshold with 10 Hz and ITI of 26 s. 1560 pulse in 40 trains at all . One train lasts 4 s.
- Total: Total of all reporting groups
Arm/Group | Verum TMS | Sham TMS | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (12.6) | 46.6 (13.7) | 44.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  Germany | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Subjective Anxiety Symptoms
Description: Change in anxiety questionaire (Agoraphobia Questionaire (AQ), subscale anxiety) from pre (baseline) to post therapy (week 4). The range of the scale is from 0 to 120. Higher values indicate higher anxiety symptoms. For the calculated changes from pre to post this means, that more negative values indicate higher symptom reductions
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verum TMS | Sham TMS
Number analyzed (Participants) | 20 | 19
units on a scale | 17.4 (15.3) | 7.3 (11.6)
Statistical Analysis 1: Comparison: Verum TMS vs Sham TMS; Test type: Superiority; p = 0.025, t-test, 1 sided

2. Primary Outcome: Subjective Anxiety in Height Situation (BAT), Differences From Pre (Baseline) to Post Therapy (Week 4)
Description: real life anxiety measurement by an behavioral approach test. Ratings on a 0-100 scale. Higher values indicate higher anxiety
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verum TMS | Sham TMS
Number analyzed (Participants) | 20 | 19
units on a scale | 25.8 (25.4) | 16.3 (13.2)
Statistical Analysis 1: Comparison: Verum TMS vs Sham TMS; Test type: Superiority; p = 0.08, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 3 month
Arm/Group | Verum TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 8/20 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum TMS (N=20) | Sham TMS (N=19)
Headache (Nervous system disorders) | 7 (7) | 1 (1)
drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes